CLINICAL TRIAL: NCT03673059
Title: A Multi-Center, Controlled Clinical Trial to Assess the Effects of Topical Lotions on Changes in the Skin Microbiome and Associations With Itch
Brief Title: Clinical Trial to Assess the Effects of Topical Lotions on Changes in the Skin Microbiome and Associations With Itch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Products Company Division of Johnson & Johnson Consumer Companies, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PS-141014142040-THCT
Record Dates: First submitted 2018-08-17; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Microbiota
Keywords: Microbiome; Eczema; Itching; Quality of life; Moisturization
MeSH Terms: conditions — Eczema; Pruritus

STUDY DESIGN:
Intervention Model Description: Subjects were randomly assigned to two groups. One group was supplied with a test product containing an OTC drug monographed ingredient for treatment of eczema and the other group was supplied with a cosmetic test product which is a standard dry skin daily moisturizer. Both groups were also provided with a cosmetic test cleanser to use in place of their normal cleanser. There was a 7-day regression period following the 14 days of product use.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OTC Eczema Moisturizer Regimen (Experimental): Subjects who were assigned to use an over-the-counter (OTC), oatmeal-containing eczema therapy moisturizing cream. The product is classified as an OTC monograph drug.
  Interventions: Drug: OTC Eczema Moisturizer Regimen
- Cosmetic Moisturizer Regimen (Experimental): Subjects who were assigned to use a non-fragranced, dry skin daily moisturizer classified as a cosmetic (i.e. non-OTC).
  Interventions: Other: Cosmetic Moisturizer Regimen

INTERVENTIONS:
Drug: OTC Eczema Moisturizer Regimen — Subjects were assigned to use an OTC, oatmeal-containing eczema therapy moisturizing cream twice daily on their face and entire body for the 14-day treatment period of the study, in place of any other moisturizers/emollients. Subjects were also provided with a mild cleanser to use in place of their normal body wash and/or soap (same cleanser as used by Group B) per their usual cleansing routine. After the 14-day treatment period, subjects discontinued use of the moisturizer for the 7-day regression period.
  Other Names: Group A
  Arms: OTC Eczema Moisturizer Regimen
Other: Cosmetic Moisturizer Regimen — Subjects were assigned to use a non-fragranced, dry skin daily moisturizer twice daily on their face and entire body for the 14-day treatment period of the study, in place of any other moisturizers/emollients. Subjects were also provided with a mild cleanser to use in place of their normal body wash and/or soap (same cleanser as used by Group A) per their usual cleansing routine. After the 14-day treatment period, subjects discontinued use of the moisturizer for the 7-day regression period.
  Other Names: Group B
  Arms: Cosmetic Moisturizer Regimen

SUMMARY:
This was a multi-center, 14-day clinical use study with a 7-day regression period, being conducted to assess the changes in the skin microbiome with two moisturizers in female and male subjects 16-50 years of age with mild to moderate eczema that experienced a recent itch flare up.

DETAILED DESCRIPTION:
In this study, subjects were divided into two groups, one group was supplied with a test product containing an over-the-counter (OTC) drug monographed ingredient for treatment of eczema. The other group was supplied with a cosmetic test product which is a standard dry skin daily moisturizer. Both groups were also provided with a cosmetic test cleanser to use in place of their normal cleanser. Subjects used the products for 14 days, followed by a 7-day regression period (no product use).

Subjects were assessed at Baseline and at Day 1, Day 3, Day 7, and Day 14 of product use. They were assessed again 7 days after stopping product use. Only the group provided with the test product containing the monograph ingredient for treatment of eczema were assessed for eczema endpoints after the Baseline visit.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate eczema, as determined by the investigator (score of 2.0-7.5 on Rajka-Langeland severity index).
* Has 1 target lesion, as determined by the investigator (score of 6-12 on Atopic Dermatitis Severity Index (ADSI) and sub-score of at least 2 on erythema and pruritus).
* Experienced a recent itch flare up and is experiencing pre-flare up symptoms at screening.
* Did not use moisturizer on the face and body for 3 days prior to screening.
* Has a score of at least 4.0 on Visual Analog Scale (VAS) Itch Assessment scale at baseline.
* Generally in good health.
* Willing to stop using all topical emollients, moisturizers, and/or other skin barrier creams and/or emulsion treatments for the eczema condition during the test period.
* Willing and able to follow all study directions, including avoiding excessive sun exposure (including tanning beds), and to commit to all follow up visits for the duration of the study.
* Completed informed consent/assent process and signed photograph release.
* Must agree to practice a medically acceptable form of birth control.

Exclusion Criteria:

* Known allergies or sensitivities to test product ingredients.
* Severe eczema.
* Using a therapeutic (over the counter or prescription) body wash that contains an active ingredient for eczema.
* Has a health condition or skin condition that the study investigator thinks could increase risk to the subject or confuse study results (e.g. immune deficiency disorders).
* Has been using that the study investigator thinks could increase risk to the subject or confuse study results (e.g. corticosteroids, immunosuppressive medications).
* Currently participating in another study.
* Subjects who have clinically active bacterial, fungal, or viral skin infections or those who are susceptible to cutaneous infections.
* Has any planned surgery and/or invasive medical procedures scheduled during the course of the study.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2016-06-13 (Actual)

PRIMARY OUTCOMES:
Microbiome Composition Changes in Lesion Skin - Baseline to Day 14 | 2 weeks
  Changes in the composition (abundance and diversity) of the microbiome communities present on the lesional skin from Baseline to Day 14. The microbiome of the skin of interest was sampled using a sterile swab, sequenced to amplify genomic regions, and analyzed using standard protocols to determine associated organisms, both known and novel, between the two time points.

SECONDARY OUTCOMES:
Microbiome Composition Changes in Lesion Skin - Baseline to Day 7 | 1 week
  Changes in the composition (abundance and diversity) of the microbiome communities present on the lesional skin from Baseline to Day 7. The microbiome of the skin of interest was sampled using a sterile swab, sequenced to amplify genomic regions, and analyzed using standard protocols to determine associated organisms, both known and novel, between the two time points.
Microbiome Composition Changes in Lesion Skin - Baseline to Day 3 | 3 days
  Changes in the composition (abundance and diversity) of the microbiome communities present on the lesional skin from Baseline to Day 3. The microbiome of the skin of interest was sampled using a sterile swab, sequenced to amplify genomic regions, and analyzed using standard protocols to determine associated organisms, both known and novel, between the two time points.
Microbiome Composition Changes in Lesion Skin - Baseline to Day 1 | 1 day
  Changes in the composition (abundance and diversity) of the microbiome communities present on the lesional skin from Baseline to Day 1. The microbiome of the skin of interest was sampled using a sterile swab, sequenced to amplify genomic regions, and analyzed using standard protocols to determine associated organisms, both known and novel, between the two time points.
Microbiome Composition Changes in Lesion Skin - Regression Baseline to Day Regression Day 7 | 1 week
  Changes in the composition (abundance and diversity) of the microbiome communities present on the lesional skin from Regression Baseline (Study Day 14) to Regression Day 7 (Study Day 21). The microbiome of the skin of interest was sampled using a sterile swab, sequenced to amplify genomic regions, and analyzed using standard protocols to determine associated organisms, both known and novel, between the two time points.
Skin pH - Change - Baseline to Day 14 | 2 weeks
  Change from baseline in pH of lesional skin at Day 14.
Skin pH - Change - Baseline to Day 7 | 1 week
  Change from baseline in pH of lesional skin at Day 7.
Skin pH - Change - Baseline to Day 3 | 3 days
  Change from baseline in pH of lesional skin at Day 3.
Skin pH - Change - Baseline to Day 1 | 1 day
  Change from baseline in pH of lesional skin at Day 1.
Skin pH - Change - Regression Baseline to Regression Day 7 | 1 week
  Change from regression baseline (Study Day 14) in pH of lesion skin at Regression Day 7 (Study Day 21).
Skin Transepidermal Water Loss (TEWL) - Change - Baseline to Day 14 | 2 weeks
  Change from baseline in TEWL of lesional skin at Day 14.
Skin Transepidermal Water Loss (TEWL) - Change - Baseline to Day 7 | 1 week
  Change from baseline in TEWL of lesional skin at Day 7.
Skin Transepidermal Water Loss (TEWL) - Change - Baseline to Day 3 | 3 days
  Change from baseline in TEWL of lesional skin at Day 3.
Skin Transepidermal Water Loss (TEWL) - Change - Baseline to Day 1 | 1 day
  Change from baseline in TEWL of lesional skin at Day 1.
Skin Transepidermal Water Loss (TEWL) - Change - Regression Baseline to Regression Day 7 | 1 week
  Change from regression baseline (Study Day 14) in TEWL of lesional skin at Regression Day 7 (Study Day 21).
Skin Hydration - Change - Baseline to Day 14 | 2 weeks
  Change from baseline in Skin Hydration via conductance of lesional skin at Day 14.
Skin Hydration - Change - Baseline to Day 7 | 1 week
  Change from baseline in Skin Hydration via conductance of lesional skin at Day 7.
Skin Hydration - Change - Baseline to Day 3 | 3 days
  Change from baseline in Skin Hydration via conductance of lesional skin at Day 3.
Skin Hydration - Change - Baseline to Day 1 | 1 day
  Change from baseline in Skin Hydration via conductance of lesional skin at Day 1.
Skin Hydration - Change - Regression Baseline (Day 14) to Regression Day 7 (Day 21) | 1 week
  Change from regression baseline (Day 14) in Skin Hydration via conductance of lesional skin at Regression Day 7 (Day 21).
Eczema Area Severity Index (EASI) - Change - Baseline to Day 14 | 2 weeks
  Change from baseline in total EASI score at Day 14. Group A only. The EASI scoring system provides a score that reflects the severity of clinical signs of eczema based on the percentage of affected area in each of 4 body regions - the head/neck, trunk, upper extremities, and lower extremities. Each body region is scored for 4 parameters: erythema, edema, excoriations, and lichenification on a 0 (none) to 3 (severe) scale. The score for these parameters is summed and then multiplied by a constant that reflects the relative body area of that body region (head/neck = 0.10; trunk = 0.30; upper extremities = 0.20, lower extremities = 0.40). The total EASI score is calculated as a sum of the scores for the 4 individual body regions. The total possible score ranges from 0 (no eczema anywhere on the body) to 72 (severest eczema symptoms on all body areas).
Eczema Area Severity Index (EASI) - Change - Baseline to Day 7 | 1 week
  Change from baseline in total EASI score at Day 7. Group A only. The EASI scoring system provides a score that reflects the severity of clinical signs of eczema based on the percentage of affected area in each of 4 body regions - the head/neck, trunk, upper extremities, and lower extremities. Each body region is scored for 4 parameters: erythema, edema, excoriations, and lichenification on a 0 (none) to 3 (severe) scale. The score for these parameters is summed and then multiplied by a constant that reflects the relative body area of that body region (head/neck = 0.10; trunk = 0.30; upper extremities = 0.20, lower extremities = 0.40). The total EASI score is calculated as a sum of the scores for the 4 individual body regions. The total possible score ranges from 0 (no eczema anywhere on the body) to 72 (severest eczema symptoms on all body areas).
Eczema Area Severity Index (EASI) - Change - Baseline to Day 3 | 3 days
  Change from baseline in total EASI score at Day 3. Group A only. The EASI scoring system provides a score that reflects the severity of clinical signs of eczema based on the percentage of affected area in each of 4 body regions - the head/neck, trunk, upper extremities, and lower extremities. Each body region is scored for 4 parameters: erythema, edema, excoriations, and lichenification on a 0 (none) to 3 (severe) scale. The score for these parameters is summed and then multiplied by a constant that reflects the relative body area of that body region (head/neck = 0.10; trunk = 0.30; upper extremities = 0.20, lower extremities = 0.40). The total EASI score is calculated as a sum of the scores for the 4 individual body regions. The total possible score ranges from 0 (no eczema anywhere on the body) to 72 (severest eczema symptoms on all body areas).
Eczema Area Severity Index (EASI) - Change - Baseline to Day 1 | 1 day
  Change from baseline in total EASI score at Day 1. Group A only. The EASI scoring system provides a score that reflects the severity of clinical signs of eczema based on the percentage of affected area in each of 4 body regions - the head/neck, trunk, upper extremities, and lower extremities. Each body region is scored for 4 parameters: erythema, edema, excoriations, and lichenification on a 0 (none) to 3 (severe) scale. The score for these parameters is summed and then multiplied by a constant that reflects the relative body area of that body region (head/neck = 0.10; trunk = 0.30; upper extremities = 0.20, lower extremities = 0.40). The total EASI score is calculated as a sum of the scores for the 4 individual body regions. The total possible score ranges from 0 (no eczema anywhere on the body) to 72 (severest eczema symptoms on all body areas).
Eczema Area Severity Index (EASI) - Change - Regression Baseline to Regression Day 7 | 1 week
  Change from regression baseline (Study Day 14) in total EASI score at Regression Day 7 (Study Day 21). Group A only. The EASI scoring system provides a score that reflects the severity of clinical signs of eczema based on the percentage of affected area in each of 4 body regions - the head/neck, trunk, upper extremities, and lower extremities. Each body region is scored for 4 parameters: erythema, edema, excoriations, and lichenification on a 0 (none) to 3 (severe) scale. The score for these parameters is summed and then multiplied by a constant that reflects the relative body area of that body region (head/neck = 0.10; trunk = 0.30; upper extremities = 0.20, lower extremities = 0.40). The total EASI score is calculated as a sum of the scores for the 4 individual body regions. The total possible score ranges from 0 (no eczema anywhere on the body) to 72 (severest eczema symptoms on all body areas).
Atopic Dermatitis Severity Index (ADSI) - Change - Baseline to Day 14 | 2 weeks
  Change from baseline in total ADSI score at Day 14. Group A only. ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, itching, exudation, excoriation, lichenification - which are each measured on a 0 (none) to 3 (scale). The total score can range from 0 (no eczema signs) to 15 (very severe eczema lesion).
Atopic Dermatitis Severity Index (ADSI) - Change - Baseline to Day 7 | 1 week
  Change from baseline in total ADSI score at Day 7. Group A only. ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, itching, exudation, excoriation, lichenification - which are each measured on a 0 (none) to 3 (scale). The total score can range from 0 (no eczema signs) to 15 (very severe eczema lesion).
Atopic Dermatitis Severity Index (ADSI) - Change - Baseline to Day 3 | 3 days
  Change from baseline in total ADSI score at Day 3. Group A only. ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, itching, exudation, excoriation, lichenification - which are each measured on a 0 (none) to 3 (scale). The total score can range from 0 (no eczema signs) to 15 (very severe eczema lesion).
Atopic Dermatitis Severity Index (ADSI) - Change - Baseline to Day 1 | 1 day
  Change from baseline in total ADSI score at Day 1. Group A only. ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, itching, exudation, excoriation, lichenification - which are each measured on a 0 (none) to 3 (scale). The total score can range from 0 (no eczema signs) to 15 (very severe eczema lesion).
Atopic Dermatitis Severity Index (ADSI) - Change - Regression Baseline to Regression Day 7 | 1 week
  Change from regression baseline (Study Day 14) in total ADSI score at Regression Day 7 (Study Day 21). Group A only. ADSI is a scoring system that reflects the severity of a target eczema lesion. The ADSI score is a sum of scores for 5 different parameters - erythema, itching, exudation, excoriation, lichenification - which are each measured on a 0 (none) to 3 (scale). The total score can range from 0 (no eczema signs) to 15 (very severe eczema lesion).

CONTACTS AND LOCATIONS:
Overall Officials: Lily Jiang, Ph.D., Principal Investigator — Thomas J. Stephens & Associates, Inc.
Locations (2):
- United States (2):
  - Thomas J. Stephens & Associates, Inc., Colorado Springs, Colorado
  - Thomas J. Stephens and Associates, Inc., Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phan NQ, Blome C, Fritz F, Gerss J, Reich A, Ebata T, Augustin M, Szepietowski JC, Stander S. Assessment of pruritus intensity: prospective study on validity and reliability of the visual analogue scale, numerical rating scale and verbal rating scale in 471 patients with chronic pruritus. Acta Derm Venereol. 2012 Sep;92(5):502-7. doi: 10.2340/00015555-1246. PMID 22170091
- [Background] Desai NS, Poindexter GB, Monthrope YM, Bendeck SE, Swerlick RA, Chen SC. A pilot quality-of-life instrument for pruritus. J Am Acad Dermatol. 2008 Aug;59(2):234-44. doi: 10.1016/j.jaad.2008.04.006. Epub 2008 Jun 11. PMID 18550210
- [Background] Lipozencic J, Wolf R. Atopic dermatitis: an update and review of the literature. Dermatol Clin. 2007 Oct;25(4):605-12, x. doi: 10.1016/j.det.2007.06.009. PMID 17903619
- [Background] Elman S, Hynan LS, Gabriel V, Mayo MJ. The 5-D itch scale: a new measure of pruritus. Br J Dermatol. 2010 Mar;162(3):587-93. doi: 10.1111/j.1365-2133.2009.09586.x. Epub 2009 Dec 1. PMID 19995367
- [Background] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Background] Rajka G, Langeland T. Grading of the severity of atopic dermatitis. Acta Derm Venereol Suppl (Stockh). 1989;144:13-4. doi: 10.2340/000155551441314. PMID 2800895
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575